CLINICAL TRIAL: NCT00194142
Title: Cytomegalovirus (CMV) Infection in Amniotic Fluid
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 803583; R01 17625-03-14
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Pregnancy Complications; Cytomegalovirus Infections
Keywords: Pregnancy; Cytomegalovirus
MeSH Terms: conditions — Pregnancy Complications; Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to determine if detection of cytomegalovirus (CMV) in amniotic fluid collected in the second trimester of pregnancy is associated with pregnancy complications such as preterm delivery or severe preeclampsia.

DETAILED DESCRIPTION:
CMV infection in adults with a normal immune system is rarely a serious event. Once a person has been infected with CMV, they may have recurrences (relapses) of the infection. If a mother is infected with the virus or relapses during pregnancy, her fetus may be at risk for infection. Unlike infection in adults, congenital infection may result in serious complications (congenital infection). The effects of fetal infection with CMV are well understood and many efforts have been made to potentially reduce the risk of congenital infection. However, the effect of CMV infection on the pregnancy itself (when the fetus is not affected by CMV) is less understood.

The incidence of CMV detection in amniotic fluid collected in the second trimester is thought to be low. However, the association between detection of CMV infection in the second trimester and ultimate pregnancy outcome is poorly described.

In this study, we plan to determine if CMV detection in amniotic fluid collected in the second trimester is associated with pregnancy complications.

ELIGIBILITY:
Inclusion Criteria:

* Women who deliver at term without pregnancy complications
* Women who deliver (preterm, less than 37 weeks of gestation) as a result of spontaneous preterm labor
* Women whose pregnancies are complicated by severe preeclampsia

Exclusion Criteria:

* Women with multi-gestational pregnancies, or whose pregnancies are complicated by a congenital malformation or chromosomal abnormality
* Women who have a medical history of hypertension (high blood pressure), diabetes, or severe renal (kidney) disease

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The purpose of this study is to determine the prevalence of Cytomegalovirus (CMV) infection in amniotic fluid specimens obtained at 16 to 18 weeks of pregnancy and to determine if CMV infection of amniotic fluid supernatant and/or amniocytes is associated with adverse obstetric outcomes. Amniotic fluid will be obtained from an already established registry. and analyzed in conjunction with a chart review under a HIPAA Waiver of Authorization.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2007-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doris Chou, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States